CLINICAL TRIAL: NCT02643875
Title: Investigation of the Effect of Short-term Orthokeratology With Increased Compression Factor on Ocular Parameters
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Collaborators: Menicon Co., Ltd. (Industry); Queensland University of Technology (Other); Aston University (Other)
Responsible Party: Principal Investigator, Pauline Cho, Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: HSEARS20151002004
Record Dates: First submitted 2015-12-28; First posted 2015-12-31 (Estimated); Results first posted 2020-09-18 (Actual); Last update posted 2020-09-18 (Actual); Status verified 2020-02

CONDITIONS: Myopic Progression
Keywords: myopia control; orthokeratology

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (2):
- Ortho-k lens with normal compression factor (Sham Comparator): The eye wears ortho-k lens with normal compression factor to achieve plano (+/- 0.25D) correction.
  Interventions: Device: Orthokeratology
- Ortho-k lenses with increased compression factor (Active Comparator): The eye wears ortho-k lenses with increased compression factor to achieve 1 diopter (+/- 0.25D) over correction.
  Interventions: Device: Orthokeratology

INTERVENTIONS:
Device: Orthokeratology — It is a kind of rigid permeable lens.

SUMMARY:
Orthokeratology (ortho-k) is a clinical technique that uses reverse geometry rigid gas permeable contact lens exerting positive pressure on the central cornea to temporary reduce refractive error. Researchers have shown that this treatment is effective for myopia control in low to high myopes, with and without astigmatism. Most designs of ortho-k lenses in the market are fitted based on the Jessen formula. The compression factor was introduced to compensate for the regression of the ortho-k effect during the no lens-wear period, so that the wearer can obtain clear distance vision throughout the day and most lens designs use a compression factor of 0.50-0.75 D. However, in a retrospective study (mixed brands of ortho-k lenses), it showed that most patients did not achieve an over-correction of 0.75 D. In order to achieve an over-correction of 0.75 D, an extra flattening power of about 1.50 D instead of 0.75 D should be be targeted. The increased compression factor is expected to increase the target reduction and it may play a role in myopic control and providing a higher successful rate in fitting ortho-k lenses.

DETAILED DESCRIPTION:
Subjects were fitted with ortho-k lenses of conventional (0.75 D) and increased (1.75 D) compression factor. The laterality of the compression factor for each subject was randomised.

Subjects were instructed and trained with proper lens handling and disinfection procedures. Lenses were given to the subjects only when they demonstrated proper techniques.

All subjects were required to attend regular follow-ups (baseline, first overnight, and weekly over one-month period). The follow-ups were scheduled (except for the first overnight which was scheduled in the early morning) at a similar time to the baseline visit (+/- 2 hours) to minimise any potential influence of diurnal variation on ocular biometrics.

Additional unscheduled visits were provided when necessary to ensure good ocular health and vision throughout the study period.

ELIGIBILITY:
Inclusion Criteria:

1. 6 to 10 years old
2. Myopia: between 0.50 D and 4.00 D in both eyes
3. Astigmatism: <1.50 D; ≤ 1.25 D for with-the-rule astigmatism (axes 180 ± 30); ≤ 0.50 D for astigmatism of other axes in both eyes
4. Anisometropia: ≤ 1.50 D
5. Symmetrical corneal topography with corneal toricity <2.00 D in both eyes
6. Agree for randomization

Exclusion Criteria:

1. Contraindications for orthokeratology wear (e.g. limbus-to-limbus corneal cylinder and dislocated corneal apex)
2. Any type of strabismus or amblyopia
3. Myopic treatment (e.g. refractive surgery and progressive lens wear for myopic control) before and during the study period
4. Rigid contact lenses (including orthokeratology lenses) experience
5. Systemic condition which might affect refractive development (for example, Down syndrome, Marfan's syndrome)
6. Ocular conditions which might affect the refractive error (for example, cataract, ptosis)
7. Poor compliance for lens wear or follow-up

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 36 (Actual)
Dates: Start 2016-02-26 (Actual); Primary Completion 2016-11-18 (Actual); Study Completion 2016-11-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pauline Cho, PhD, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- The Hong Kong Polytechnic University, Hong Kong, China

REFERENCES:
- [Background] Cho P, Cheung SW, Edwards M. The longitudinal orthokeratology research in children (LORIC) in Hong Kong: a pilot study on refractive changes and myopic control. Curr Eye Res. 2005 Jan;30(1):71-80. doi: 10.1080/02713680590907256. PMID 15875367
- [Background] Cho P, Cheung SW. Retardation of myopia in Orthokeratology (ROMIO) study: a 2-year randomized clinical trial. Invest Ophthalmol Vis Sci. 2012 Oct 11;53(11):7077-85. doi: 10.1167/iovs.12-10565. PMID 22969068
- [Background] Chen C, Cheung SW, Cho P. Myopia control using toric orthokeratology (TO-SEE study). Invest Ophthalmol Vis Sci. 2013 Oct 3;54(10):6510-7. doi: 10.1167/iovs.13-12527. PMID 24003088
- [Background] Chan B, Cho P, Mountford J. The validity of the Jessen formula in overnight orthokeratology: a retrospective study. Ophthalmic Physiol Opt. 2008 May;28(3):265-8. doi: 10.1111/j.1475-1313.2008.00545.x. PMID 18426426
- [Result] Wan K, Lau JK, Cheung SW, Cho P. Refractive and corneal responses of young myopic children to short-term orthokeratology treatment with different compression factors. Cont Lens Anterior Eye. 2020 Feb;43(1):65-72. doi: 10.1016/j.clae.2019.10.134. Epub 2019 Nov 6. PMID 31704093
- [Result] Lau JK, Vincent SJ, Cheung SW, Cho P. The influence of orthokeratology compression factor on ocular higher-order aberrations. Clin Exp Optom. 2020 Jan;103(1):123-128. doi: 10.1111/cxo.12933. Epub 2019 Jul 1. PMID 31264269
- [Result] Lau JK, Wan K, Cheung SW, Vincent SJ, Cho P. Weekly Changes in Axial Length and Choroidal Thickness in Children During and Following Orthokeratology Treatment With Different Compression Factors. Transl Vis Sci Technol. 2019 Jul 23;8(4):9. doi: 10.1167/tvst.8.4.9. eCollection 2019 Jul. PMID 31360614

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All subjects who passed the inclusion and exclusion criteria at the baseline visit would be assigned to the treatment for each eye according to the randomization log.
Units Other Than Participants: eyes
Groups:
- Orthokeratology Lenses With Different Compression Factors: Orthokeratology lenses with different compression factors (one eye with 0.75 D and the fellow eye with 1.75 D) were randomly assigned to each subject.
Period: Overall Study
Arm/Group | Orthokeratology Lenses With Different Compression Factors
Started | 36; 72 eyes
Received 0.75 | 36; 36 eyes
Received 1.75 D | 36; 36 eyes
Completed | 28; 56 eyes
Not Completed | 8; 16 eyes

BASELINE CHARACTERISTICS:
Population: Data of subjects who completed the study were reported
Units Other Than Participants: eyes
Arm/Group | Orthokeratology Lenses With Different Compression Factors
Number analyzed (Participants) | 28
Number analyzed (eyes) | 56
Age, Continuous [Mean (Full Range); unit: years] | 9.3 [7.8 to 11.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 12
Spherical equivalent refraction [Mean (Standard Deviation); unit: D] — Maximum plus for maximum visual acuity was used as the criterion for subjective refraction.
  Spherical equivalent refraction was calculated by adding the sum of the sphere power with half of the cylinder power. Population: Orthokeratology lenses with different compression factors (one eye with 0.75 D and the fellow eye with 1.75 D) were randomly assigned to each subject.
  D
    number analyzed (eyes) | 28
    Conventional compression factor (0.75 D) | 2.12 (0.94)
    Increased compression factor (1.75 D) | 2.09 (0.97)

OUTCOME MEASURES:

1. Primary Outcome: Changes in Spherical Equivalent Refraction
Description: Maximum plus for maximum visual acuity was used as the criterion for subjective refraction.
  Spherical equivalent refraction was calculated by adding the sum of the sphere power with half of the cylinder power.
Time Frame: baseline and one month
Population: Orthokeratology lenses with different compression factors (one eye with 0.75 D and the fellow eye with 1.75 D) were randomly assigned to each subject.
Measure: Mean (Standard Deviation); unit: D
Units Other Than Participants: eyes
Arm/Group | Orthokeratology Lenses With Different Compression Factors
Number analyzed (Participants) | 28
Number analyzed (eyes) | 56
D
  Conventional compression factor (0.75 D): number analyzed (eyes) | 28
  Conventional compression factor (0.75 D) | 2.31 (0.88)
  Increased compression factor (1.75 D): number analyzed (eyes) | 28
  Increased compression factor (1.75 D) | 2.52 (0.85)

2. Secondary Outcome: Changes in Subfoveal Choroidal Thickness
Description: The subfoveal choroidal thickness was determined as the thickness between the outer retinal pigment epithelium/Bruch's membrane complex and the inner chorioscleral interface.
Time Frame: baseline and one month
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: um
Units Other Than Participants: eyes
Arm/Group | Orthokeratology Lenses With Different Compression Factors
Number analyzed (Participants) | 28
Number analyzed (eyes) | 56
um
  Conventional compression factor (0.75 D): number analyzed (eyes) | 28
  Conventional compression factor (0.75 D) | -1 (30)
  Increased compression factor (1.75 D): number analyzed (eyes) | 28
  Increased compression factor (1.75 D) | -6 (30)

3. Secondary Outcome: Changes in Higher Order Aberrations
Description: Ocular higher order aberrations were measured using Shack-Hartmann aberrometer. The wavefront data was fitted with a sixth order Zernike polynomial over a 5-mm pupil size.
Time Frame: baseline and one month
Population: as for outcome 1
Measure: Mean (Standard Error); unit: um
Units Other Than Participants: eyes
Arm/Group | Orthokeratology Lenses With Different Compression Factors
Number analyzed (Participants) | 28
Number analyzed (eyes) | 56
um
  Conventional compression factor (0.75 D): number analyzed (eyes) | 28
  Conventional compression factor (0.75 D) | 0.2830 (0.03)
  Increased compression factor (1.75 D): number analyzed (eyes) | 28
  Increased compression factor (1.75 D) | 0.1870 (0.03)

ADVERSE EVENTS:
Time Frame: one month
Groups:
- Conventional Compression Factor (0.75 D): Orthokeratology lenses with conventional compression factor (0.75 D) were randomly assigned to one eye of each subject.
- Increased Compression Factor (1.75 D): Orthokeratology lenses with increased compression factor (1.75 D) were randomly assigned to the fellow eye of each subject.
Arm/Group | Conventional Compression Factor (0.75 D) | Increased Compression Factor (1.75 D)
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/28
Other Adverse Events (participants affected / at risk) | 0/28 | 0/28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes